CLINICAL TRIAL: NCT04279405
Title: A Phase 1b Study to Assess the Safety and Efficacy of YY-20394 in Subjects With Recurrent and/or Refractory B-cell Hematologic Malignancies
Brief Title: A Phase Ib Study of YY-20394 in Participants With B-cell Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-007
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): treatment with YY-20394 will be continued until tumor progression or development of unacceptable toxicity.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — YY-20394 80mg tablet administered orally once daily

SUMMARY:
Protocol YY-20394-007 is a phase1 open-label, single-arm, multi-centre study to assess the safety and efficacy of YY-20394 in participants with relapse and/or refractory B cell malignant hematological tumor. eligible participants will initiate oral therapy with YY-20394 at a starting dose of 80mg taken once per day. treatment with YY-20394 can continue in compliant participants as long as the study is still ongoing and the participants appear to benefiting from treatment with acceptable safety.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed relapse and/or refractory B cell hematologic malignancies(Excluding follicular lymphoma)
* prior treatment with ≥1 prior standard anti-tumor regimens and 2 courses of treatments at least
* eastern cooperative oncology group performance status of 0 to 2
* life expectancy of at least 3 months
* presence of >1.5cm radiographically measurable lymphadenopathy or extranodal lymphoid malignancy, and legibility in two vertical directions
* acceptable organ functions
* discontinuation of all other antitumor therapies before the first drug dose administration
* for men and women of childbearing potential, willingness to abstain from sexual intercourse or employ an effective method of contraception during the study drug administration and follow-up six periods
* willingness and ability to provide written informed consent and to comply with the protocol requirements

Exclusion Criteria:

* prior therapy with PI3K-delta inhibitors（except the intolerable subjects）
* the dosage of steroid hormone(predisone equivalent) was greater than 20mg/d, and lasted for more than 14 days
* medical condition of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditional that may hamper compliance and/or absorption of the investigational product
* concurrent drugs which maybe prolong the QT during the study period
* subjects with central nervous system metastasis
* Prior or current medical condition of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc
* active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* known history of chronic active hepatitis B infection, chronic active hepatitis C
* known history of immunodeficiency, including HIV positive test, other acquired or congenital immunodeficiency disorders, organ transplantation or allogeneic bone marrow transplantation
* autologous hematopoietic stem cell transplantation was received within 90 days before the first dose administration
* prior or ongoing heart disease, including: angina pectoris, clinically significant arrhythmia, myocardial infarction, heart failure, and any other heart disease judged by the researchers not eligible to the study
* pregnancy or breastfeeding
* prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant or impair the assessment of study results
* receiving granulocyte colony-stimulating factor(GCSF) or blood transfusion within seven days before screening
* history of a non-lymphoma malignancy except for adequately treated local basal cell carcinoma of the skin and cervical carcinoma in situ
* subjects, in the opinion of the the Investigator, who are unsuitable to participate in the study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse events evaluated by NCI CTCAE V5.0 | Throughout the study for approximately 2 years
  incidence of adverse events and associated dose of YY-20394
Overall response rate | Throughout the study for approximately 2 years
  the percentage of participants achieving a complete response or partial response
disease control rate | Throughout the study for approximately 2 years
  the percentage of participants achieving a complete response or partial response or stable disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, China